CLINICAL TRIAL: NCT04436159
Title: Partial Versus Total Fundoplication in the Surgical Repair of Para-esophageal Hernia. Results of a Randomized Clinical Trial
Brief Title: Partial Versus Total Fundoplication in the Surgical Repair of Para-esophageal Hernia.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska University Hospital (Other)
Collaborators: Ersta Hospital, Sweden (Other)
Responsible Party: Principal Investigator, Lars Lundell, Professor, Karolinska University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2008/179-31
Record Dates: First submitted 2020-06-16; First posted 2020-06-17 (Actual); Last update posted 2021-09-02 (Actual); Status verified 2021-08

CONDITIONS: Paraesophageal Hernia; Gastro Esophageal Reflux
Keywords: Nissen fundoplication; Toupet fundoplication; crural repair; Quality of Life
MeSH Terms: conditions — Hernia, Hiatal; Gastroesophageal Reflux

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nissen fundoplication (Active Comparator): Addition of 360 fundoplication after crural closure
  Interventions: Procedure: Addition of 360 fundoplication after crural closure
- Toupet fundoplication (Active Comparator): Addition of 180 posterior fundoplication after crural closure
  Interventions: Procedure: Addition of 180 posterior fundoplication after crural closure

INTERVENTIONS:
Procedure: Addition of 360 fundoplication after crural closure — A total fundoplication was constructed in which the right and left part of the wrap was brought together in front of, and slightly to the right of the esophagus, and sutured with three interrupted stitches of 2-0 unabsorbable sutures from the GEJ and cranially to attain a length between the top and bottom sutures of at the most 2 cm. At least one wrap suture included the esophageal muscle-wall.
  Arms: Nissen fundoplication
Procedure: Addition of 180 posterior fundoplication after crural closure — The wrap was pulled dorsally around the distal part of the esophagus and GEJ, which was encircled approximately 180-200 degrees. First, the wrap was anchored with Gore-tex sutures, dorsally to the left crus with 3 sutures and then to the right crus with another 3 sutures.
  Finally, the wrap was completed with 3-4 sutures, between the edges of the wrap and the right and left side of the esophageal wall, respectively.
  Arms: Toupet fundoplication

SUMMARY:
Short-term follow up after surgery of para-esophageal hernia comparing two different types of fundoplication

DETAILED DESCRIPTION:
Laparoscopic para-esophageal hernia (PEH) repair has been established as a safe and effective treatment for symptomatic patients. Today, most surgeons agree that a fundoplication should be included in the hiatal reconstruction in order to reduce the risk of postoperative gastroesophageal reflux and hernia recurrence. However, what type of wrap that should be recommend is yet to be determined.

One might argue that the overall durability and effectiveness of a partial fundoplication in the control of reflux might be less reliable than a total wrap, but on the contrary, the latter carries the risk of inducing a pseudoachalasia similar situation in PEH patients.

We therefore designed a double blind randomized clinical trial in which patients with symptomatic paraesophageal hernia to receive either a posterior partial (Toupet) or total (Nissen) fundoplication after hernia reduction and crural repair.

Six months follow up with questionnaires, 24-hour pH monitoring and radiology after surgery of para-esophageal hernia with addition of total fundoplication vs posterial partial fundoplication.

Dysphagia Scores; Ogilvie dysphagia score and Watson dysphagia score. Quality of Life; SF-36: physical and mental component scores.

Time points: 1, 3 and 6 months after surgery

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing acute or elective surgery for symptomatic PEH at Ersta Hospital and Karolinska University Hospital

Exclusion Criteria:

* age below 18 years
* axial sliding hiatal hernia only (type I)
* missing informed consent
* previous hiatal hernia surgery
* American Society of Anesthesiologists (ASA) score IV or above
* achalasia
* Zollinger-Ellison syndrome
* malignant tumor
* inability or unwillingness to complete questionnaires

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2018-09 (Actual); Study Completion 2018-09 (Actual)

PRIMARY OUTCOMES:
Ogilvie dysphagia score | 6 months
  The Ogilvie dysphagia score is a 5-graded scale 0-4 defined as follows: '0', ability to eat ordinary diet; '1', ability to swallow solid food; '2', ability to swallow semisolids; '3', ability to swallow liquids; '4', total inability to swallow .

SECONDARY OUTCOMES:
intra-and postoperative courses | 6 mohths
  Peri and postoperative complications.
length of hospital stay | 6 months
  postoperative length of hospital stay
Watson dysphagia score | 6 months
  Watson dysphagia score is a validated instrument for benign dysphagia where the patient is asked whether he/she always, sometimes or never has difficulty swallowing nine different groups of liquid and food items.
  This gives a score ranging from zero to 45, where 45 represents the worst possible dysphagia.
Acid reflux control | 6 months
  24-hour pH monitoring
Quality of Life (SF-36) | 6 months
  The Swedish version of this validated global questionnaire is presented as physical and mental summary component scores (PCS and MCS, respectively). Each subscale scores reaches a value of at the most 100, where higher values reflect better health status.
Radiology | 6 months
  Radiologically verified recurrent hiatal hernia

CONTACTS AND LOCATIONS:
Overall Officials: Lars Lundell, professor, Principal Investigator — Karolinska Institutet
Locations (1):
- Ersta Hospital, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Analatos A, Lindblad M, Ansorge C, Lundell L, Thorell A, Hakanson BS. Total versus partial posterior fundoplication in the surgical repair of para-oesophageal hernias: randomized clinical trial. BJS Open. 2022 May 2;6(3):zrac034. doi: 10.1093/bjsopen/zrac034. PMID 35511051